CLINICAL TRIAL: NCT01674959
Title: Phase II Study of Postoperative Intensity-modulated Radiotherapy (IMRT) Combined With Capecitabine for Stage II/III Gastric Cancer Patients
Brief Title: Postoperative IMRT Combined With Capecitabine for Advanced Gastric Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Attending doctor of Dept. radiation oncology, Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011 CH-GI-024
Record Dates: First submitted 2012-08-26; First posted 2012-08-29 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; radiation; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- concurrent chemoradiation (Experimental): • Radiation: concurrent chemoradiotherapy Postoperative radiotherapy regimen: Therapy plan system was formulated by Computed tomographic (CT) simulation. Radiation was delivered with 6MV photons. Radiotherapy consisted of 4500 cGy of radiation at 180 cGy per day, five days per week for five weeks, to the tumor bed, to the margins of resection or the stoma, to the regional nodes. Protection of spinal cord, heart, liver and kidney should be considered.
  Postoperative current chemotherapy regimen: capecitabine( 1,600 mg/m2 per day for 5 weeks).
  Interventions: Radiation: concurrent chemoradiation

INTERVENTIONS:
Radiation: concurrent chemoradiation — postoperative Intensity-modulated radiotherapy (IMRT) combined with capecitabine for high risk gastric cancer patients Radiation: concurrent chemoradiotherapy Postoperative radiotherapy regimen: Therapy plan system was formulated by Computed tomographic (CT) simulation. Radiation was delivered with 6MV photons. Radiotherapy consisted of 4500 cGy of radiation at 180 cGy per day, five days per week for five weeks, to the tumor bed, to the margins of resection or the stoma, to the regional nodes. Protection of spinal cord, heart, liver and kidney should be considered.
  Postoperative chemotherapy regimen: capecitabine( 1,600 mg/m2 per day for 5 weeks).

SUMMARY:
Radiation therapy plus concurrent chemotherapy has been demonstrated a significant improvement in overall and disease-free survival according to Intergroup Trial 0116 in patients with gastric cancer after surgical complete resection. Advantage of application of IMRT has been shown in planning comparison studies for postoperative gastric patients. So the investigators designed the trial to see safety and efficacy of postoperative concurrent chemoradiotherapy of capecitabine combined with IMRT for stage II/II gastric cancer.

DETAILED DESCRIPTION:
In Intergroup 0116, only 64% patients in concurrent chemoradiation group completed treatment as planed, but in recently reported ARTIST trial, capecitabine was admitted to concurrent with radiotherapy,patients who completed treatment as planed in concurrent group reach high as 80%. IMRT is an advanced radiotherapy technology which allows high conformal dose distribution to Planing Tumor Volume (PTV) and low dose to organ at risk. The purpose of this study is to evaluate feasibility and efficacy of concurrent IMRT combined with capecitabine for the treatment of gastric cancer patients after D1/2 surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative histologically confirmed advanced adenocarcinoma of the stomach or the gastroesophageal junction.
2. Age of 18 to 75, Karnofsky score higher than 70.
3. Postoperative histologically conformed metastasis in perigastric lymph nodes and/or tumor invasion to muscularis propria or subserosa, without positive incisal margin. Stage II/III(AJCC 7th).
4. No severe functional damage of major organ, normal blood cell, normal liver and kidney function.
5. No clinical findings of distant metastasis.
6. Predictive survival time longer than 6 months.

   -

Exclusion Criteria:

1. Peritoneal carcinomatosis, as diagnosed by mandatory laparoscopy or distant metastasis
2. Concurrent treatment with other experimental drugs or other anti-cancer therapy, or treatment within a clinical trial within 30 days prior to trial entry
3. Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, no myocardial infarction within the last 12 months, unstable angina pectoris, or significant arrhythmia)
4. Active or uncontrolled infection.
5. Definitive contraindications for the use of corticosteroids as premedication
6. Prior systemic (chemo- or targeted) treatment. Prior radiotherapy to the upper abdomen
7. Any contraindication to treatment with cetuximab, capecitabine or cisplatin
8. Previous malignancy within 5 years, with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
9. Known hypersensitivity against any of the study drugs ( capecitabine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
feasibility of concurrent IMRT combined with capecitabine for the treatment of gastric cancer patients | 3 months after concurrent chemoradiation
  feasibility of concurrent IMRT combined with capecitabine is defined as toxicities (CTC-AE 3.0) and rate of patients complete concurrent chemoradiation according to protocol.

SECONDARY OUTCOMES:
efficacy of concurrent IMRT combined with capecitabine for the treatment of gastric cancer patients | 3 years after concurrent chemoradiation
  efficacy of concurrent IMRT combined with capecitabine for the treatment of gastric cancer patients in this trial is defined as 3-year overall survival and 3-year relapse free survival.

CONTACTS AND LOCATIONS:
Overall Officials: jing jin, professor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Dept of Radiation oncology, Cancer Hospital , Chinese Academy of Medical Science, Beijing, Beijing Municipality, China